CLINICAL TRIAL: NCT02110628
Title: Jejunal Pouch for Postoperative Quality of Life Following Roux-en-Y Reconstruction of Radical Total Gastrectomy: a Multicenter Randomized Controlled Trial (WCGCC-1202)
Brief Title: Roux-en-Y vs. Roux-en-Y+ Pouch for D2 Total Gastrectomy
Acronym: WCGCC-1202
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCGCC-1202
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer; Roux-en-y Anastomosis Site; Gastric Anastomosis (Site); Quality of Life; Complication
Keywords: total gastrectomy; pouch; roux-en-y; quality of life
MeSH Terms: conditions — Stomach Neoplasms | interventions — Anastomosis, Roux-en-Y

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y+Pouch Group (Experimental): Abdominal approach D2 total gastrectomy with Roux-en-Y+Pouch anastomosis. Roux-en-Y+Pouch anastomosis: closed the stump of duodenum, cut off the jejunum from the 20cm of Treitz ligament, pouch reconstruction a J pouch with a length of 15 cm was constructed by connecting the 2 Jejunal lumina, œsophago-P type jejunum Storage bag anastomosis (duct-to-duct / duct-to-duct, before the colon/after the colon), jejunum - jejunum anastomosis (duct-to-duct / duct-to-duct), the distance between anastomotic were 40cm-60cm.
  Interventions: Procedure: Roux-en-Y+Pouch anastomosis
- Roux-en-Y group (Experimental): Abdominal approach D2 total gastrectomy with Roux-en-Y anastomosis. Roux-en-Y anastomosis : closed the stump of duodenum, cut off the jejunum from the 20cm of Treitz ligament, œsophago-jejunal anastomosis (duct-to-duct / duct-to-duct, before the colon/after the colon), jejunum - jejunum anastomosis (duct-to-duct / duct-to-duct), the distance between anastomotic were 40cm-60cm
  Interventions: Procedure: Roux-en-Y anastomosis

INTERVENTIONS:
Procedure: Roux-en-Y anastomosis — Roux-en-Y anastomosis
  Arms: Roux-en-Y group
Procedure: Roux-en-Y+Pouch anastomosis — Roux-en-Y+Pouch anastomosis
  Arms: Roux-en-Y+Pouch Group

SUMMARY:
Gastric is one of the most prevalence digestive malignance tumors in China. Radical resection of primary tumors and combine with dissection of regional lymph-nodes is acknowledged by surgeons all over the world. Nowadays, in order to improve the quality of life, controversies still exist to the reconstruction methods of total gastrectomy. Although roux-en-y anastomosis is the most common method adopted after total gastrectomy for it is an easily and safety method reconstruction method, but some problems still need us to solve, such as little food reserves, less food intake per meal and fast gastric emptying. These problems significantly affect the patients' quality of life after surgery. Roux-en-Y+Jejunal pouch anastomosis is newly born method can significant increase the volume to improve postoperative quality of life have been proven by some little sample size randomized control trail With the improvement of the gastric cancer surgery, this study proposed by prospective randomized controlled clinical trials aimed to comparing quality of life after traditional Roux-en-Y type and Roux-en-Y+ Jejunal pouch type anastomosis for radical total gastrectomy. Quality of life was evaluated according to the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ)-C30 and QLQ-STO22. Quality of life will conducted in the 3 months, 6 months, 9 months, 12 months, 24 months, 36 months after gastrectomy.

DETAILED DESCRIPTION:
Consecutive patients in each participant units and satisfied with inclusion/exclusion criteria will be informed the details, right, responsibility possible benefit and potential risks when after join in this study. Those patients who agree and sign informed consent document will randomized, consecutive case series sampling.

All the patients in the study and finished sampling would and must be recorded in the Western China Gastric Cancer Collaboration database and assign to corresponding treatment group.

Randomization allocation

After intraoperative exploration and predictively D2 radical (R0) total gastrectomy is possible to be performed, then assigned randomly to each subject on a 1:1 basis to either the Roux-en-Y+Pouch group or the Roux-en-Y group.

Surgical treatment

Surgical approach: open total gastrectomy. Surgical treatment method: Radical total gastrectomy (R0); D2 lymph-node dissection (No.1, 2, 3, 4sa, 4sb, 4d, 5, 6, 7, 8a, 9, 10, 11p, 11d, 12a,19,20); Abscission pneumogastric nerve trunk.

Reconstruction method:

Group A (Roux-en-Y type): closed the stump of duodenum, cut off the jejunum from the 20cm of Treitz ligament, esophagojejunal anastomosis (duct-to-duct / duct-to-duct, before the colon/after the colon), jejunum - jejunum anastomosis (duct-to-duct / duct-to-duct), the distance between anastomotic were 40cm-60cm; Group B (Roux-en-Y+Pouch type): closed the stump of duodenum, cut off the jejunum from the 20cm of Treitz ligament, pouch reconstruction a J pouch with a length of 15 cm was constructed by connecting the 2 Jejunal lumina, œsophago-P type jejunum Storage bag anastomosis (duct-to-duct / duct-to-duct, before the colon/after the colon), jejunum - jejunum anastomosis (duct-to-duct / duct-to-duct), the distance between anastomotic were 40cm-60cm

Quality control of surgery:

All the surgical treatments will be performed by member of Western China Gastric Cancer Collaboration. Quality supervision within groups to avoid the bias.

Intraoperative photograph after the lymphadenectomy and the reconstruction of the digestive tract is essential.

Follow-up and Database

Follow-up programming:

Postoperative follow-up and assessment will be performed by specially researchers arrange by each units and blind to randomize allocation; Postoperative long term follow-up will be conducted in 3 months, 6 months, 9 months, 12 months, 24 months, 36 months after gastrectomy; Face to face interview is necessary and the postoperative quality of life questionnaire is done by the patients themselves.

Management of the database:

The design of this study database was responsible for the leading units; Each cases of this study should and must have a uniform case reported form, include demographic data, operation data, pathological information and Postoperative quality of life evaluation; A file included in the Case Report Form (CRF) was record follow-up information last to three years after surgery.

Lost follow-up:

Three years lost follow-up rates should below 10%. Lost follow-up rate will reported in final reports, and cases of lost follow-up will take the intention-to-treat (ITT) method to analysis.

Statistics analysis The measurement data strictly obey normal distribution are presented as means (±SD) and compared with single factor analysis of variance.

The measurement data do not obey normal distribution are presented as median and compared with Wilcoxon test.

Categorical data are presented percentage and compared with the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed gastric adenocarcinoma, and predictively feasible of total gastrectomy;
2. Predictively resectable diseases, either early or locally advanced gastric cancer, of preoperative staging Japanese Gastric Cancer Association (JGCA) 14th Edition cT1N0M0-T4aN3M0, I-IIIb, except T4b;
3. Age: 18-75 years;
4. Without serious disease;
5. WHO performance score < 2;
6. No limit to sexual and race;
7. Informed consent required

Exclusion Criteria:

1. Primary lesion cannot be resected in the pattern of transabdominal total gastrectomy, but for Whipple's procedure, or combined organ resection or with a transthoracic approach surgery;
2. Patients with other gastric malignant diseases, such as lymphoma and stromal tumors etc.
3. Patients suffering from malignant diseases before the study;
4. Patients with other severe comorbidities and cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe chronic obstructive pulmonary disease (COPD), chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc.
5. Performed emergency operation due to bleeding or perforation;
6. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
7. Not the radical surgery, but with tumor residual (R1 or R2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2014-08; Primary Completion 2019-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative quality of life | 3 years
  Postoperative quality of life is evaluated by the EORTC QLQ-C30 and the EORTC QLQ-STO22

SECONDARY OUTCOMES:
Intraoperative morbidity and mortality | Intraoperative
Postoperative morbidity and mortality | within the first 30 days after surgery
Change of the postoperative body weight | 3 years
  Evaluation the change of the body weigh

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D., Principal Investigator — West China Hospital
Locations (9):
- China (9):
  - Southwest Hospital, the Third Military Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Union Hospital, Tongji Medical College, Wuhan, Hubei
  - First Affiliated Hospital of Xi'an Jiaotong University School of Medicine, Xian, Shanxi
  - Tangdu Hospital, Fourth Military Medical University, Xian, Shanxi
  - Xijing hospital, Fourth Military Medical University, Xian, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming medical University, Kunming, Yunnan

REFERENCES:
- [Derived] Hu J, Zhang W, Western China Gastric Cancer Collaboration C. [Experience and present situation of Western China Gastric Cancer Collaboration]. Zhonghua Wei Chang Wai Ke Za Zhi. 2017 Mar 25;20(3):247-250. Chinese. PMID 28338153
- See also: homepage of West China Hospital, Sichuan University — http://www.cd120.com